CLINICAL TRIAL: NCT06022276
Title: An Open ,Single Arm, Prospective and Basket Clinical Study of Nimotuzumab in the Treatment of EGFR-amplified Advanced Pan Solid Tumors (Lung/Esophageal/Gastric/Pancreatic /Colorectal / Head and Neck Cervical)
Brief Title: Nimotuzumab for EGFR-amplified Advanced Pan Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nimotuzumab for Pan-cancer
Record Dates: First submitted 2023-08-19; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; EGFR Amplification
Keywords: Solid Tumor; Nimotuzumab; EGFR
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy or combination therapy based on Nimotuzumab (Experimental): Nitozumab injection 400mg/cycle, every 21 days/cycle, until disease progression, intolerable toxicity or death, or subject decision to withdraw from the study.The molecular testing results of the patient are analyzed and interpreted by the MTB team, and appropriate combination therapy(Nitozumab+) strategies are proposed based on the patient's previous treatment history, physical condition, drug accessibility, and economic status.
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nitozumab injection 400mg/cycle, every 21 days/cycle, until disease progression, intolerable toxicity or death, or subject decision to withdraw from the study.The molecular testing results of the patient are analyzed and interpreted by the MTB team, and appropriate combination therapy(Nitozumab+) strategies are proposed based on the patient's previous treatment history, physical condition, drug accessibility, and economic status.

SUMMARY:
To evaluate the efficacy and safety of nimotuzumab in the treatment of EGFR-amplified advanced pan solid tumors (Lung/Esophageal/Gastric/Pancreatic /Colorectal / Head and neck Cervical).

DETAILED DESCRIPTION:
Nimotuzumab is a EGFR monoclonal antibody. This clinical trial is to study the effect and safety of Nimotuzumab for EGFR-amplified advanced pan solid tumors (Lung/Esophageal/Gastric/Pancreatic /Colorectal / Head and neck Cervical) in the real world. The amplification of the patient's EGFR can be determined by tissue-next-generation sequencing (NGS), Liquid-NGS, or fluorescence in situ hybridization (FISH) . EGFR-amplified status identified in any Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. EGFR-amplified status also was assessed for pathogenicity in each case by MTB.Meanwhile, the molecular testing results of the patient are analyzed and interpreted by the MTB team, and appropriate combination therapy(Nitozumab+) strategies are proposed based on the patient's previous treatment history, physical condition, drug accessibility, and economic status. In addition, exploring molecular markers that can predict the efficacy of Nimotuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal cancer, gastric cancer, pancreatic cancer, colorectal cancer (left colorectal cancer), head and neck cancer (including oral cancer, oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer, nasopharyngeal cancer, oropharyngeal cancer must be p16 negative: p16 ≥ 70% is positive), cervical cancer, local recurrence or with distant metastasis. Patients with known EGFR amplification and standard treatment depletion or inability to tolerate standard treatment and disease progression. Allow patients with stable symptoms of brain metastasis to be enrolled.
2. Age 18-80 years old, both male and female. Expected life>3 months.
3. According to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1), there should be at least one measurable lesion that has not undergone local treatment such as radiotherapy (lesions located within the previous radiotherapy area, if confirmed to have progressed and meet the RECIST 1.1 criteria, can also be selected as target lesions).
4. It has been confirmed through NGS testing that EGFR amplification exists simultaneously (all cancer species).
5. ECOG: 0-2.
6. Expected survival time ≥ 12 weeks.
7. If the main organs function normally, they meet the following standards:

(1) Blood routine examination: a. HB ≥ 90g/L;b. ANC ≥ 1.5 × 10^9/L;c. PLT ≥ 80 × 10^9/L.

(2) Biochemical examination: a. ALB ≥ 30g/L;b. ALT and AST ≤ 2.5ULN. If there is liver metastasis, ALT and AST ≤ 5ULN; c. TBIL ≤ 1.5ULN; d. Plasma Cr ≤ 1.5ULN or creatinine clearance rate (CCr) ≥ 60ml/min.

8. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study. Within 7 days prior to enrollment in the study, the serum or urine pregnancy test was negative and must be a non-lactating patient. Men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

9. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion criteria:

1. The patient has any active autoimmune disease or autoimmune disease (For example, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism. patients with vitiligo. asthma that has completely relieved in childhood and does not require any intervention in adulthood can be included. asthma that requires medical intervention with bronchodilators cannot be included).
2. The patient is currently using systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day of prednisone or other therapeutic hormones) and continues to use it within 2 weeks before enrollment.
3. Previously received treatment with EGFR monoclonal antibodies or EGFR tyrosine kinase inhibitors.
4. Patients with any severe and/or uncontrollable diseases, including:

   Patients with poor blood pressure control (systolic blood pressure ≥ 150mm Hg or diastolic blood pressure ≥ 100 mmHg). Suffering from grade I or above myocardial ischemia or infarction, arrhythmia (including QT interval ≥ 480ms), and grade I cardiac dysfunction. Active or uncontrollable serious infections. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 10^4 copies/ml or 2000IU/ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analytical method).
5. Patients whose imaging shows that the tumor has invaded important blood vessels or who have been determined by the researchers to be highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies.
6. Pregnant or lactating women.
7. Patients with other malignant tumors within 5 years (excluding cured skin basal cell carcinoma and cervical carcinoma in situ).
8. Patients who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders.
9. Patients who have participated in clinical trials of other drugs within four weeks.
10. Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS2/PFS1 | Through study completion, an expected average of 1 year
  The progression free survival (PFS1) after the most recent treatment before enrollment is defined as the progression of the disease from the most recent treatment before enrollment.The progression free survival period (PFS2) after enrollment is defined as the time from matched targeted therapy or unmatched therapy to disease progression or death.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | Through study completion, an expected average of 1 year
  The proportion of patients whose tumor volume is reduced to 30% and can be maintained for more than 4 weeks,Based on RECIST criteria v1.1.
Progression-free Survival(PFS) | The last subject completes at least 24 weeks of follow-up (or disease progression).
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST criteria v1.1.
Disease control rate(DCR) | Through study completion,an expected average of 1 year
  The DCR was defined as SD, PR or CR according to RECIST criteria v1.1.
Overall survival(OS) | Through study completion, an expected average of 2 years.
  The time from the patient receiving treatment to the death of the patient for any reason,OS evaluated according to RECIST v1.1.
Duration of Response(DOR) | Through study completion, an expected average of 1 year
  Duration of Response,from the first time the evaluation results meet CR or PR criteria to the observation of PD or death.
Adverse events(AEs） | Through study completion, an expected average of 2 years.
  Include Treatment emerge adverse events, treatment related adverse events and serious adverse events,AEs evaluated according to NCI-CTCAE v5.0.
Quality of Life(QoL) | Through study completion, an expected average of 2 years.
  The Quality of Life scale was used to represent patients' satisfaction with quality of life to evaluate the changes in QOL of patients before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: HaiTao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China